CLINICAL TRIAL: NCT04053244
Title: A Single-Centre, Open-Label Trial of Therapist-Assisted Internet-Based Cognitive Behaviour Therapy for Cardiac Patients With Depression
Brief Title: Internet-based Cognitive Behavioural Therapy for Cardiac Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Martha Mackay, Cardiac Clinical Nurse Specialist, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-01695
Record Dates: First submitted 2019-08-07; First posted 2019-08-12 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Depression; Cardiovascular Diseases
Keywords: iCBT; cardiac event; cognitive behavioural therapy; depression
MeSH Terms: conditions — Depression; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A Single-Centre, Open-Label Trial of Therapist-Assisted Internet-Based Cognitive Behaviour Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): all participants will be assigned to the treatment, consisting of therapist-assisted iCBT.
  Interventions: Behavioral: internet-based cognitive behavioural therapy

INTERVENTIONS:
Behavioral: internet-based cognitive behavioural therapy — Designed for general clinical use (but not specifically cardiac patients), it consists of 5 online modules outlining cognitive-behavioural skills for depression, completed over 7-8 weeks. The participants will be guided step-wise through the modules by the therapist. Participants can work more or less at their own pace, but are expected to proceed to the next module within 1-2 weeks. Because the content is identical for each participant, fidelity to the web-based component of the intervention is ensured.

SUMMARY:
Our overall objective is to evaluate the efficacy of therapist-assisted, internet-based cognitive-behavioural therapy (iCBT) for depressed cardiac patients with respect to clinical outcomes, and the feasibility of the program. Our primary outcome will be depression severity; secondary outcomes will be hospitalization for a cardiac cause, recurrent myocardial infarction or revascularization. The study will inform a proposal to incorporate iCBT into the resources routinely available to cardiac patients following hospitalization for a cardiac event.

DETAILED DESCRIPTION:
We are planning we are planning a single-arm, open label trial to evaluate the feasibility, acceptability and efficacy of iCBT among persistently depressed cardiac patients. Cardiac patients will be recruited from inpatient units in a university-affiliated hospital and screened for depression at 4 and possibly 8 or 12 weeks following discharge. Eligible patients will be enrolled in the iCBT program.Data regarding the primary outcome, improvement in depression severity, will be collected at completion of the intervention and at 8 weeks after completion. In addition to depression severity data, we will also obtain other data related to clinical feasibility, such as treatment adherence and the acceptability of the intervention to patients. Self-reported rates of hospital readmission or emergency visits for a cardiac cause will also be tracked.

ELIGIBILITY:
Inclusion Criteria:

* admitted to one of study units with any cardiac diagnosis OR cardiac procedure on this admission
* able to speak and read English
* able to provide informed consent and participate in therapy
* access to and ability to use a computer with internet access.

Between 4 and 12 weeks after discharge, consenting participants will be required to meet a further inclusion criterion of:

• current depressive symptoms of at least mild severity on 2 successive assessments, 4 weeks apart or a single assessment of mild symptoms at 12 weeks post-discharge.

Exclusion Criteria:

Applied at screening (and criteria 1 and 2 reapplied before enrolment):

1. active suicidal ideation (since this requires immediate referral for intense psychiatric care)
2. previous suicide attempt
3. currently undergoing psychotherapy for depression
4. receiving antidepressant medication that has been initiated or adjusted within previous 3 months
5. concurrent psychiatric disorder, other than anxiety;
6. self-reported substance misuse within past 6 months
7. concurrent terminal illness
8. clinical status interfering with ability to independently engage in iCBT.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Depression Severity | baseline, completion of treatment (average of 12 weeks), study completion (treatment completion + 8 weeks)
  change in severity of depression as measured by Patient Health Questionnaire-9

SECONDARY OUTCOMES:
major adverse cardiac events | completion of treatment, average of 8 weeks
  death, myocardial infarction, revascularization, hospitalization for a cardiac cause
Treatment Satisfaction Questionnaire | completion of treatment, average of 8 weeks
  participants' satisfaction with treatment
Web-Based Program Usability Questionnaire | completion of treatment, average of 8 weeks
  participants' experience with using the web-based program

CONTACTS AND LOCATIONS:
Overall Officials: Martha H Mackay, PhD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
We would share all of our de-identified, individual-level data with any credentialed researcher.
Supporting Information: Study Protocol, SAP, ICF